CLINICAL TRIAL: NCT02734524
Title: A Clinical Research of NK Cell Infusion Combined With Chemotherapy in the Treatment of Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Shiqi Li, Researcher of Biotherapy Center, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMMU-BTC-004
Record Dates: First submitted 2015-11-08; First posted 2016-04-12 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Natural killer cells; NSCLC; NCT; Combined therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Taxes; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NK infusion+chemotherapy (Experimental): Treatment includes four cycles. For each cycle: Taxol and carboplatin will be given at the first week. Lymphodepletion will be conducted at the second week. Autologous NK cells will be infused at the third week. Each cycle includes four weeks.
  Interventions: Biological: NK cells; Drug: Taxol; Drug: Carboplatin
- chemotherapy (Active Comparator): Receive the same taxol and carboplatin in experimental arm without NK cell infusion.
  Interventions: Drug: Taxol; Drug: Carboplatin

INTERVENTIONS:
Biological: NK cells — Natural killer cell infusion is an intervention between two arms. Dosage of infused cell >1×10^9，q28d*4
  Other Names: natural killer cell infusion
  Arms: NK infusion+chemotherapy
Drug: Taxol — 135-175mg/m2,q28d*4
  Other Names: TAX
Drug: Carboplatin — AUC=5,q28d*4
  Other Names: Cis-platinum

SUMMARY:
The main purpose of this study is to explore if the combination of autologous NK cell infusion and chemotherapy can increase the therapeutic efficiency in the treatment of non-small cell lung cancer compared with chemotherapy alone.

DETAILED DESCRIPTION:
Natural killer cells play an important role in the anti-tumor process mediated by innate immunity. However, past researches showed dissatisfactory clinical outcome in clinicaltrials using autologous NK cell infusion alone. With the expectation that the combination of autologous NK cell infusion and chemotherapy may increase the therapeutic efficiency of chemotherapy alone in cancer treatment, the investigators design and conduct this randomized controlled trial in the treatment of non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Non-small cell lung cancer must be diagnosed by pathology and staged as ⅢB or Ⅳ with 2009-UICC TNM staging system and operation is excluded due to medical reasons or patient's will.
2. According to Response Evaluation Criteria in Solid Tumors(RECIST), at least one measurable or evaluable nidus can be detected by chest CT.
3. ECOG score 0-1.
4. Gender is not limited, age from 18 years to 75 years.
5. Patients are expected to survive for more than 3 months by their physicians at the time of enrollment.
6. Mental state is evaluated as normal.
7. Adequate cardiac function(LVEF≥40%, tested within one month) without heart diseases.
8. Hepatic and renal function were normal, biochemical criterion must meet the requests below: white blood cell count≥2.5×10^9/L，platelet count≥100×10^9/L，hemoglobin≥90g/L, serum bilirubin≤2 upper limit of normal(ULN), AST and ALT≤2 ULN(AST, ALT≤5ULN under hepatic metastases), Bun≤2 ULN, serum creatinine≤2 ULN.
9. No other serious illnesses(e.g.,autoimmune disease, immunodeficiency, ect.).
10. Ability to give informed consent.
11. No other malignancies diagnosed.
12. Patients volunteer to participate in the research.

Exclusion Criteria:

Subjects meeting any of the following criteria are not eligible for participation in the study:

1. Frequent infection history and recent infection is uncontrolled.
2. Patients with concomitant genetic syndrome: patients with Down syndrome, Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known bone marrow failure syndrome
3. Concurrent use of systemic steroids or chronic use of immunosuppressant medications. Recent or current use of inhaled steroids is not exclusionary. For additional details regarding use of steroid and immunosuppressant medications.
4. Pregnancy and nursing females.
5. HIV infection.
6. Active hepatitis B or active hepatitis C.
7. Participation in a prior investigational study within 4 weeks prior to enrollment or longer if required by local regulation. Participation in non-therapeutic research studies is allowed.
8. Class III/IV cardiovascular disability according to the New York Heart Association Classification.
9. Patients with a known history or prior diagnosis of other serious immunologic, malignant or inflammatory disease.
10. Other situations we think not eligible for participation in the research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants responding to treatment | 4 months
  Response evaluation of treatment with chest CT scan is assessed by RECIST 1.1

SECONDARY OUTCOMES:
Progress free survival(PFS) time | 2 years
Overall survival time | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Qian, MD, PhD, Study Chair — Biotherapy Center of Southwest Hospital
Locations (1):
- Southwest Hospital of Third Millitary Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided